CLINICAL TRIAL: NCT06726252
Title: A Prospective, Multicenter, Self-controlled Clinical Trial to Validate Optical Ultrasonic Flow Ratio (OUFR) Based on Intravascular Imaging
Brief Title: Prospective, Multicenter, Self-controlled Clinical Trial to Validate Optical Ultrasonic Flow Ratio (OUFR)
Acronym: OUFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Peking University Third Hospital (Other); Panovision (Unknown); Capital Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Jining Medical University (Other); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yu Bo, Director, cardiology department, the 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Optical Ultrasonic Flow Ratio
Record Dates: First submitted 2024-11-12; First posted 2024-12-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Fractional Flow Reserve; Coronary Artery Disease
Keywords: FFR; IVUS; OCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Validation of OUFR using wire-based FFR measurement as the gold standard (Experimental): Participants undoing anticipated percutaneous coronary intervention will be performed wire-based FFR measurement and intravascular imaging, including IVUS and integrated OCT-IVUS using a single catheter, to assess the sensitivity, specificity and oter performance measures of OUFR, using wire-based FFR as the gold standard.
  Interventions: Device: FFR measurement and intravascular imaging

INTERVENTIONS:
Device: FFR measurement and intravascular imaging — Participants undoing anticipated percutaneous coronary intervention will be performed wire-based FFR measurement, and intravascular imaging, including IVUS and integrated OCT-IVUS using a single cathete to assess the accurary of OUFR, using wire-based FFR measurement as the gold standard.

SUMMARY:
The objective of is study is to validate a novel computational Fractional Flow Reserve (FFR) index method, termed Optical Ultrasonic Flow Ratio (OUFR), based on intravascular imaging including intravascular optical coherence tomography (OCT) and intravascular ultrasound (IVUS), using wire-based FFR as the gold standard. This is a prospective, multi-center, self-controlled clinical trial involving at least four medical centers and recruiting at least 114 subjects based on statistical power analysis.

Participants undoing anticipated percutaneous coronary intervention will be performed:

1. Wire-based FFR measurement
2. Intravascular imaging, including IVUS and integrated OCT-IVUS using a single catheter.

The primary endpoint is to assess patient-level sensitivity, specificity of OUFR computed based on OCT; (2) OUFR based on IVUS, and OUFR based on both OCT and IVUS, using wire-based FFR measurement as the gold standard.

DETAILED DESCRIPTION:
The objective of this study is to verify a novel computational Fractional Flow Reserve (FFR) index method, termed Optical Ultrasonic Flow Ratio (OUFR), based on intravascular imaging including intravascular optical coherence tomography (OCT) and intravascular ultrasound (IVUS). This is a prospective, multi-center, self-controlled clinical trial involving at least four medical centers to verify OUFR using wire-based FFR measurement as the gold standard.

Subjects: At least 114 subjects will be recruited based on statistical power analysis.

The primary inclusion criteria include: (1) At least 18 years old; (2) Anticipate to be performed percutaneous coronary intervention (PCI); (3) Can sustain FFR measurement, IVUS and OCT imaging; (4) Understand the objective of this study, and sign informed consent form voluntarily. (5) The pullback of intravascular imaging covers the FFR measurement site and the entire stenotic lesion, and the OCT and IVUS images are of sufficient quality for OUFR analysis.

Specific exclusion criteria include: (1) Women with pregnancy or anticipate to be pregnant within 6 months; (2) Participated in other clinical studies within 3 months; (3) Had acute coronary syndromes within 30 days; (4) Heart failure (NYHA III or NYHA IV, or left ventricular ejection fraction<30%); (5) Abnormal levels of cTnI or cTnT within 72 hours of the procedure; (6) Had coronary artery bypass grafting surgery; (7) Diagnosed as bacteremia or septicemia; (8) Diagnosed as coronary artery spasm; (9) Clinically significant abnormal coagulation function; (10) Clinically significant abnormal liver or kidney function; (11) Clinically significant hemodynamic disorders or coma; (12) Allergic to contrast or have other potential risks due to allergy; (13) Presence of clinical unstable conditions, including acute chest pain, cardiogenic shock, unstable blood pressure (e.g. systolic pressure < 90mmHg), severe congestive heart failure or acute pulmonary edema; (14) Presence of other medical conditions not suitable for participating in this clinical study, such as complex congenital heart disease, myocardial bridge, long QT syndrome (LQTS), severe asthma, severe chronic obstructive pulmonary disease (COPD), or COPD with a dependency on bronchodilator, or with other severe infection or acute diseases; (15) Reference vessel diameter outside the range of 2.0-4.0mm by angiography, and diameter stenosis outside the range of 30%-90%; (16) Lesions associated with left main or coronary ostium, target vessel with severe tortuosity or calcified lesions, coronary total occlusion, diffuse lesions; (17) Target vessel with thrombus or dissection confirmed by angiography; (18) Target vessel with previous stenting; (19) Target vessel with the minimum lumen diameter < 1.1mm; (20) TIMI flow grade≤2; (21) Balloon predilatation before FFR wire measurement or intravascular imaging; (22) FFR wire or intravascular imaging catheter cannot pass the stenotic lesion; (23) Unable to observe maximal hyperemia during FFR measurement or failure to obtain FFR data; (24) Intravascular imaging failure due to the damage of imaging catheters or insufficient blood clearance, or operational factors; (25) Presence of vasospasm or injury during imaging; (24) Other reasons identified by investigators that preclude the subjects from participating in the study.

Main intervantional procedure: (1) For subjects meeting all the inclusion criteria, obtain the informed consent; (2) Apply exclusion criteria based on medical history and conditions; (3) Perform coronary angiography; (4) Perform FFR measurement using the pressure wire from Abbott (IL, USA); (5) Perform intravascular imaging with the C1-1 catheter from Panovision (Beijing, China) to obtain IVUS and integrated OCT-IVUS pullback images; (6) Apply exclusion criteria based on angiography, FFR and intravascular imaging, if necessary; (7) Collect data from all centers and send the data to an independent Corelab from the lead institution for OUFR computation and statistical analysis.

Primary endpoints: With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate patient-level sensitivity, specificity of (1) OUFR computed based on OCT (OUFRo); (2) OUFR based on IVUS (OUFRi); and (3) OUFR based on both OCT and IVUS (OUFRoi).

Secondary endpoints: With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate (1) Vessel-level sensitivity and specificity of OUFRo, OUFRi and OUFRoi; (2) Patient-level accuracy of OUFRo, OUFRi and OUFRoi; (3) Patient and vessel level positive predictive value (PPV), negative predictive value (NPV) and area under the ROC curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Anticipate to be performed percutaneous coronary intervention (PCI)
* Can sustain FFR measurement, IVUS and OCT imaging
* Understand the objective of this study, and sign informed consent form voluntarily
* The pullback of intravascular imaging covers the FFR measurement site and the entire stenotic lesion, and the OCT and IVUS images are of sufficient quality for OUFR analysis

Exclusion Criteria:

* Women with pregnancy or anticipate to be pregnant within 6 months
* Participated in other clinical studies within 3 months
* Had acute coronary syndromes within 30 days
* Heart failure (NYHA III or NYHA IV, or left ventricular ejection fraction<30%)
* Abnormal levels of cTnI or cTnT within 72 hours of the procedure
* Had coronary artery bypass grafting surgery
* Diagnosed as bacteremia or septicemia
* Diagnosed as coronary artery spasm
* Clinically significant abnormal coagulation function
* Clinically significant abnormal liver or kidney function
* Clinically significant hemodynamic disorders or coma
* Allergic to contrast or have other potential risks due to allergy
* Presence of clinical unstable conditions, including acute chest pain, cardiogenic shock, unstable blood pressure (e.g. systolic pressure < 90mmHg), severe congestive heart failure or acute pulmonary edema
* Presence of other medical conditions not suitable for participating in this clinical study, such as complex congenital heart disease, myocardial bridge, long QT syndrome (LQTS), severe asthma, severe chronic obstructive pulmonary disease (COPD), or COPD with a dependency on bronchodilator, or with other severe infection or acute diseases
* Reference vessel diameter outside the range of 2.0-4.0mm by angiography, and diameter stenosis outside the range of 30%-90%
* Lesions associated with left main or coronary ostium, target vessel with severe tortuosity or calcified lesions, coronary total occlusion, diffuse lesions
* Target vessel with thrombus or dissection confirmed by angiography
* Target vessel with previous stenting
* Target vessel with the minimum lumen diameter < 1.1mm
* TIMI flow grade≤2
* Balloon predilatation before FFR wire measurement or intravascular imaging
* FFR wire or intravascular imaging catheter cannot pass the stenotic lesion
* Unable to observe maximal hyperemia during FFR measurement or failure to obtain FFR data
* Intravascular imaging failure due to the damage of imaging catheters or insufficient blood clearance, or operational factors
* Presence of vasospasm or injury during imaging
* Other reasons identified by investigators that preclude the subjects from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Patient-level sensitivity and specificity | "From enrollment to the end of data analysis, up to 12 months
  With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate patient-level sensitivity, specificity of (1) OUFR computed based on OCT (OUFRo); (2) OUFR based on IVUS (OUFRi); and (3) OUFR based on both OCT and IVUS (OUFRoi).

SECONDARY OUTCOMES:
Vessel-level sensitivity and specificity of OUFR | "From enrollment to the end of data analysis, up to 12 months
  With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate (1) Vessel-level sensitivity and specificity of OUFRo, OUFRi and OUFRoi
Patient-level accuracy of OUFR | From enrollment to the end of data analysis, up to 12 months
  With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate patient-level accuracy of OUFRo, OUFRi and OUFRoi
Patient and vessel level positive predictive value (PPV), negative predictive value (NPV) and area under the ROC curve (AUC) | From enrollment to the end of data analysis, up to 12 months
  With wire-based FFR measurement as the gold standard, using FFR=0.8 as the diagnostic threshold (FFR≤0.8: positive, FFR>0.8: negative), evaluate patient and vessel level positive predictive value (PPV), negative predictive value (NPV) and area under the ROC curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Harbin Medical University, Harbin, Heilongjiang
  - Jining Medical University, Jining, Shandong

IPD SHARING:
Plan to Share IPD: No
Due to patient data privacy and the national and institutional regulations, IPD will not be shared.

REFERENCES:
- [Background] Huang J, Emori H, Ding D, Kubo T, Yu W, Huang P, Zhang S, Gutierrez-Chico JL, Akasaka T, Wijns W, Tu S. Diagnostic performance of intracoronary optical coherence tomography-based versus angiography-based fractional flow reserve for the evaluation of coronary lesions. EuroIntervention. 2020 Sep 18;16(7):568-576. doi: 10.4244/EIJ-D-19-01034. PMID 31951207
- [Background] Jia H, Zhao C, Yu H, Wang Z, Liu H, Xu M, Hu S, Li L, He L, Weng Z, Qin Y, Xu Y, Zeng M, Su X, Liu B, Hou J, Yu B. Clinical performance of a novel hybrid IVUS-OCT system: a multicentre, randomised, non-inferiority trial (PANOVISION). EuroIntervention. 2023 Jul 17;19(4):e318-e320. doi: 10.4244/EIJ-D-22-01058. No abstract available. PMID 37057604
- [Background] Yu W, Huang J, Jia D, Chen S, Raffel OC, Ding D, Tian F, Kan J, Zhang S, Yan F, Chen Y, Bezerra HG, Wijns W, Tu S. Diagnostic accuracy of intracoronary optical coherence tomography-derived fractional flow reserve for assessment of coronary stenosis severity. EuroIntervention. 2019 Jun 20;15(2):189-197. doi: 10.4244/EIJ-D-19-00182. PMID 31147309